CLINICAL TRIAL: NCT01072695
Title: A Phase 2, Randomized, Open-Label Trial of GS-9256 Plus GS-9190 Alone and in Combination With Ribavirin for 28 Days in Treatment Naïve Subjects With Chronic Genotype 1 Hepatitis C Virus Infection (Protocol No. GS-US-196-0112)
Brief Title: Efficacy and Safety Study of GS-9256 and GS-9190 Alone and in Combination With Ribavirin for 28 Days in Patients With Chronic Hepatitis C Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-196-0112
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: HCV Infection
Keywords: Hepatitis C; HCV; GS-9256; GS-9190; Genotype 1
MeSH Terms: conditions — Hepatitis C | interventions — GS-9256; tegobuvir; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: GS-9256; Drug: GS-9190
- Arm 2 (Experimental)
  Interventions: Drug: GS-9256; Drug: GS-9190; Drug: Ribavirin
- Arm 3 (Experimental)
  Interventions: Drug: GS-9256; Drug: GS-9190; Drug: Ribavirin; Drug: Peginterferon alfa-2a

INTERVENTIONS:
Drug: GS-9256 — 75 mg BID x 28 days
Drug: GS-9190 — 40 mg BID x 28 days
Drug: Ribavirin — 1000-1200 mg/day given BID
  Other Names: COPEGUS
  Arms: Arm 2; Arm 3
Drug: Peginterferon alfa-2a — 180 ug q week
  Other Names: Pegasys
  Arms: Arm 3

SUMMARY:
This a phase 2, randomized, open-label trial of GS-9256 plus GS-9190, two oral anti HCV drugs, for 28 days with and without ribavirin (RIBA) and with pegylated interferon (PEG)/RIBA in adults with chronic Hepatitis C virus (HCV). In Part A, approximately thirty (30) subjects 18-70 years of age who meet study entry criteria will be randomized (in other words, selected at random, like flipping a coin) to one of the two treatment groups (GS-9256 plus GS-9190 or GS-9256 plus GS-9190 plus RIBA). In Part B, an additional fifteen (15) subjects will receive 75 mg GS-9256 BID plus 40 mg GS-9190 BID in combination with PEG/RIBA. After the 28-day treatment period, subjects will receive PEG/RIBA as standard of care (SOC).

Following randomization, subjects will return for a Baseline (Day 1) visit, at which time study medication will be dispensed and subjects will enter a 28 day treatment phase. During the treatment phase, subjects will receive oral study drugs twice daily for 28 days and PEG once weekly for Part B. Subjects then receive PEG/RIBA as local SOC starting on Day 28 (not provided as part of the study). Following completion of the 28-day treatment phase, subjects will be followed for approximately 72 weeks.

DETAILED DESCRIPTION:
GS-9256 (an HCV NS3 protease inhibitor) plus GS-9190 (non-nucleoside HCV NS5B inhibitor) will be administered for 28 days with and without RIBA (weight-based dosing) and with PEG/RIBA in treatment-naïve subjects with chronic genotype 1 HCV infection. In Part A, thirty (30) subjects with genotype 1 will be randomized to 75 mg GS-9256 BID plus 40 mg GS-9190 BID or 75 mg GS-9256 BID plus 40 mg GS-9190 BID plus RIBA 1000-1200 mg/day for 28 days. In Part B, an additional fifteen (15) subjects with genotype 1 will receive 75 mg GS-9256 BID plus 40 mg GS-9190 BID in combination with PEG/RIBA for 28 days. After the 28-day treatment period, subjects will receive PEG/RIBA as standard of care (SOC).

In Part A, for any subjects meeting pre-defined, individual, virologic criteria, PEG/RIBA standard of care will be started prior to Day 28.

Both PEG and RIBA will be administered at their currently approved dosages for treatment of HCV infection in accordance with appropriate labeling. Subjects will be monitored for safety (including ECG monitoring), antiviral activity, pharmacokinetics, and resistance 2-3 times weekly through Day 28.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects, ages 18-70
* Willing able to provide informed consent
* BMI between 18 and 36 kg/m2 (inclusive)
* Chronic HCV infection, genotype 1
* HCV RNA >/= 3 log, but < 7.2 log10 IU/ml at screen
* Liver biopsy, FibroTest, or FibroScan indicating absence of cirrhosis
* HCV treatment naïve with imminent plans to start treatment with PEG/RIBA
* QTcF </= 450 msec at screen
* ALT, AST, GGT < 5 X ULN at the screening visit
* Creatinine clearance >= 50 mL/min
* Absolute neutrophil count >= 1500/mm3
* Hemoglobin >/= 12 g/dL (female), >/= 13 g/dL (male)
* Males agree to use of effective contraception and refrain from sperm donation
* Able to comply with dosing instructions and study visits
* Of generally good health

Exclusion Criteria:

* Females of child-bearing potential or males with female partners who are pregnant or planning to become pregnant
* Infection with other HCV genotype or multiple HCV genotypes
* Poorly controlled diabetes
* Hemoglobinopathy or known retinal disease
* History of sarcoidosis or invasive malignancy
* Untreated or significant psychiatric illness
* Co-infection with hepatitis B virus or human immunodeficiency virus
* Chronic use of systemic immunosuppressive agents
* Autoimmune disorders
* Severe COPD
* History of significant cardiac disease
* Known cirrhosis
* Non-HCV chronic liver disease
* Transplantation
* Suspicion of hepatocellular carcinoma
* Bilirubin above the normal range or Gilbert's syndrome
* Decompensated liver disease
* Clinically significant illness
* GI disease that could interfere with absorption
* Acute porphyria
* Current excessive alcohol ingestion, averaging > 3 drinks/day for females and > 4 drinks/day for males or current binge drinking
* Positive urine drug screen
* History of difficult blood collection
* Significant recent blood loss
* Prohibited medications, including H2 antagonists, investigational agents
* Restricted fruits, fruit juices
* Hypersensitivity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-02; Primary Completion 2010-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving rapid virologic response (RVR) | Day 28
AEs, physical examination and clinical laboratory test findings, vital signs, ECGs | Throughout first six weeks of study

SECONDARY OUTCOMES:
Plasma pharmacokinetics | Throughout Day 28
Viral resistance | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Juan Betular, Study Director — Gilead Sciences
Locations (10):
- Brussels, Belgium
- France (3):
  - Clichy
  - La Tronche
  - Paris
- Germany (5):
  - Düsseldorf
  - Frankfurt
  - Hamburg
  - Hanover
  - Würzburg
- London, United Kingdom